CLINICAL TRIAL: NCT05832736
Title: Robotic Hemi-Prostatectomy With Urethral Preservation in Low and Intermediate Risk Monolateral Prostate Cancer: a Prospective Idea, Development, Exploration, Assessment and Long-term Follow-up (I.D.E.A.L.) Trial
Brief Title: Robotic Hemi-Prostatectomy With Urethral Preservation in Low and Intermediate Risk Monolateral Prostate Cancer
Acronym: RETURN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione del Piemonte per l'Oncologia (Other)
Responsible Party: Principal Investigator, Francesco Porpiglia, Prof., Fondazione del Piemonte per l'Oncologia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRCC 15/2023
Record Dates: First submitted 2023-04-03; First posted 2023-04-27 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with unilateral prostate cancer (Experimental): Patients with unilateral prostate cancer
  Interventions: Procedure: Robotic hemi-prostatectomy with urethral preservation

INTERVENTIONS:
Procedure: Robotic hemi-prostatectomy with urethral preservation — Robotic hemi-prostatectomy with urethral preservation
  Other Names: Partial prostatectomy

SUMMARY:
On the basis of the now consolidated literature and clinical experience of focal therapies, the execution of partial prostatectomy/hemiprostatectomy with robot-assisted laparoscopic technique can be proposed in a well-selected cohort of patients.

The hypothesis is that with this technique it is possible to achieve excellent levels of disease control, in terms of positive surgical margins (PSM) and biochemical recurrence of the disease (BCR), against a minimal impact as regards postoperative functional outcomes (continence and sexual power).

ELIGIBILITY:
Inclusion Criteria:

* Signature of the informed consent and consent to the use of personal data
* Prostate Specific Antigen (PSA) < 20 ng/mL
* Unilateral organ-confined disease on MRI (performed according to ESUR recommendations and reported according to PiRads V.2) or PET-PSMA (performed according to the recommendations of the EANM and reported according to "EANM standardized reporting guidelines v1.0 for PSMA-PET")
* Histological diagnosis of acinar-type prostate cancer unilateral on target biopsy and/or standard biopsy with ISUP < 3 and ipsilateral on imaging investigations
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1
* Life expectancy ≥ 5 years
* Availability of the patient's pre-operative clinical data
* Patients must be available to carry out the follow-up visits defined by the protocol
* Absence of retroperitoneal, lymph nodal, bone or visceral metastatic lesions
* Patients eligible for robot-assisted radical prostatectomy

Exclusion Criteria:

* Special histotypes of prostate cancer
* Patients with PSA > 20 ng/ml at diagnosis
* Impossibility to perform MRI (with pacemakers, claustrophobia…) or PET-PSMA
* Previous prostate surgery (TURP, adenomectomy)
* Concomitant treatment with other antineoplastic drugs including investigational endocrine therapies
* Serious underlying disease or uncontrolled medical condition including active and uncontrolled infections
* Patients with dementia or psychiatric illness that limit compliance with study requirements or that could prevent understanding and/or signing the informed consent.

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-04-12 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the robotic hemiprostatectomy technique | Baseline
  Evaluate the feasibility of the robotic hemiprostatectomy technique in both a preclinical and clinical setting as ratio between the number of hemiprostatectomies completed and the total number of prostatectomies performed

SECONDARY OUTCOMES:
Safety of the robotic hemiprostatectomy technique | 30 days
  Evaluate the safety of the robotic hemiprostatectomy technique in terms of intra and post-operative complications using the Clavien-Dindo classification.
  The Clavien-Dindo classification evaluates severity of complications in 5 groups:
  * Grade I: Any deviation from the normal postoperative course without the need for pharmacological treatment or surgical, endoscopic and radiological interventions;
  * Grade II: Requiring pharmacological treatment with drugs other than such allowed for grade I complications;
  * Grade III: Requiring surgical, endoscopic or radiological intervention (IIIa: Intervention not under general anesthesia; IIIb: Intervention under general anesthesia);
  * Grade IV Life-threatening complication requiring IC/ICU-management (IVa: single organ dysfunction; IVb: multiorgan dysfunction);
  * Grade V: Death of a patient.
Positive Surgical Margins (PSMs) rate | 30 days
  Evaluate the oncological efficacy in terms of Positive Surgical Margins (PSMs) at the final histological examination as rate between cases with Positive Surgical Margins over the total of the specimens analyzed by pathologists.
Biochemical Recurrence (BCR) rate | 5 years
  Evaluate the oncological efficacy in terms of Biochemical Recurrence (BCR) during the follow-up period as rate between patients with BCR over the total of patients in the study group.
  The BCR is any rise in the blood level of PSA (prostate-specific antigen) in prostate cancer patients after treatment with surgery or radiation.
Urinary continence after surgery | 5 years
  Evaluate the functional outcomes in terms of urinary continence during the follow-up period.
  The urinary continence will be assessed by the net weight of urine collected in the pad over 24 hours (Pad test).
  This outcome will be shown by the mont after the surgery in which the patient reach the complete continence defined as no urine loss at the Pad test.
Potency recovery after surgery | 5 years
  Evaluate the functional outcomes in terms of potency recovery during the follow-up period.
  The potency recovery will be assessed by the International Index of Erectile Function - 5 (IIEF-5) test. This test will be collected every follow-up visit and results will be shown as progression of the IIEF-5 during the 5 years after the surgery.
  The IIEF-5 contains 5 items and uses the sum scores and cutoff points to categorize the severity of the erectile dysfunction. This scale ranges from 5 points (severe erectile dysfunction) to 25 points (no erectile dysfunction).

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Porpiglia, Principal Investigator — Fondazione del Piemonte per l'Oncologia
Locations (1):
- Fondazione del Piemonte per l'Oncologia, Candiolo, TO, Italy